CLINICAL TRIAL: NCT05730634
Title: The Effect of Statin Treatment on Arterial Wall Inflammation in Patients With Diabetes Mellitus as Assessed With 68Ga-DOTATATE PET-CT
Brief Title: The Effect of Statin Treatment on Arterial Wall Inflammation as Assessed With 68Ga-DOTATATE PET-CT
Acronym: CARAMEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Nordin Hanssen, Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL65001.018.18
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2; Vascular Inflammation
Keywords: statin; dotatate; vascular inflammation; type 2 diabetes mellitus; pet/ct; positron emmission tomography
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Atorvastatin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Atorvastatin 40mg once daily.
  Interventions: Drug: Atorvastatin 40 Mg Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin 40 Mg Oral Tablet — Atorvastatin 40mg once daily for three months

SUMMARY:
To study the effect of atorvastatin treatment on vascular uptake of 68Ga-DOTATATE in patients with Type 2 Diabetes.

DETAILED DESCRIPTION:
Well controlled patients with type 2 diabetes, who are statin naïve, will undergo atorvastatin treatment. Before and after treatment, patients will undergo a 68Ga-DOTATATE PET/CT, to evaluate the effect of treatment on vascular inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50 years and older
2. Diagnosed with diabetes mellitus type 2 and using oral glucose lowering therapy, insulin or combined glucose lowering therapy.
3. Not on statin therapy or willing to stop with current statin therapy for 6 weeks prior to visit 2.
4. HbA1c values below 65 mmol/L.
5. Patients with "stable" diabetes mellitus, i.e. no changes in type of glucose lowering therapy and / or dosage of oral glucose lowering therapy in the past three months. No more than 20% change in dosage of insulin therapy (short and long acting) in the last three months.

Exclusion Criteria:

1. History of cardiovascular disease (previous CV-event (MI / stroke) or known coronary artery disease (including acute coronary syndrome).
2. History of chronic kidney disease stage 3b - 5, defined as a CKD-EPI value of < 45 ml/min/1,73m2
3. Malignant diseases or any clinically significant medical condition that could interfere with the conduct of the study in the opinion of the investigator.
4. Chronic or recent (< 1 month) infections and/or clinical signs of acute infection.
5. History of auto-immune diseases.
6. Standard contra-indications to 68Ga-Dotatate PET, and CT based on physicians experience and current practices.
7. Inability or unwillingness to comply with the protocol requirements, or deemed by investigator to be unfit for the study.
8. Planned radiation exposure in the next year due to participation in a research project with radiation exposure or for clinical reasons.
9. Elevated liver enzymes (> 2 ULN of liver transaminases), acute liver failure or known liver disease.
10. Prior medium to severe statin-related side effects or statin related hypersensitivity, i.e.

    (severe) muscle pains with and/or without myopathy .
11. The concomitant use of statin contra-indicated drugs, including the use of CYP3A4 inhibitors (i.e. erytromycin, dilthiazem, amiodaron, verapamil, fluconazole, ciclosporin, stiripentol, itraconazol, ketoconazol, voriconazol, posaconazol, clarithromycin, ..), systemic use of fusidic acid and ciclosporin.
12. Any contra-indications to the use of statins.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
DOTATATE coronary arteries | 3 months
  Change in DOTATATE TBRmax coronary arteries after atorvastatin therapy

SECONDARY OUTCOMES:
Change in splenic/bone marrow DOTATATE signal | 3 month
  The secondary objective of this study is to assess the feasibility to measure splenic and bone-marrow inflammatory activity with 68Ga-Dotatate PET-CT in patients with diabetes mellitus, expressed as SUVmax

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oostveen RF, Kaiser Y, Stahle MR, Nurmohamed NS, Tzolos E, Dweck MR, Kroon J, Murphy AJ, Dey D, Slomka PJ, Verberne HJ, Stroes ESG, Hanssen NMJ. Atorvastatin lowers 68Ga-DOTATATE uptake in coronary arteries, bone marrow and spleen in individuals with type 2 diabetes. Diabetologia. 2023 Nov;66(11):2164-2169. doi: 10.1007/s00125-023-05990-9. Epub 2023 Aug 15. PMID 37581619